CLINICAL TRIAL: NCT00945802
Title: A Multi-Center, Randomized, Double-Masked Clinical Study Evaluating the Efficacy Of FST-201 (Dexamethasone 0.1%) Otic Suspension (Foresight Biotherapeutics, Inc.) Vs. Ciprodex (Ciprofloxacin 0.3%, Dexamethasone 0.1%) Otic Suspension (Alcon Laboratories, Inc.) in Subjects With Acute Otitis Externa
Brief Title: FST-201 In The Treatment of Acute Otitis Externa
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FST201-AOE-02
Record Dates: First submitted 2009-07-23; First posted 2009-07-24 (Estimated); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Acute Otitis Externa
MeSH Terms: interventions — Dexamethasone; Ciprofloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- FST-201 (dexamethasone 0.1%) Otic Suspension (Experimental)
  Interventions: Drug: FST-201 (dexamethasone 0.1%) Otic Suspension
- ciprofloxacin 0.3%, dexamethasone 0.1% (Active Comparator)
  Interventions: Drug: ciprofloxacin 0.3%, dexamethasone 0.1%

INTERVENTIONS:
Drug: FST-201 (dexamethasone 0.1%) Otic Suspension — Instill four drops two times a day
  Arms: FST-201 (dexamethasone 0.1%) Otic Suspension
Drug: ciprofloxacin 0.3%, dexamethasone 0.1% — Instill four drops two times a day
  Other Names: Ciprodex
  Arms: ciprofloxacin 0.3%, dexamethasone 0.1%

SUMMARY:
The objective of this study is to evaluate the efficacy of FST-201 compared to Ciprodex in the treatment of acute otitis externa. This trial is designed to enable filing of a New Drug Application in support of FST-201 for the indication of acute otitis externa.

ELIGIBILITY:
Inclusion Criteria:

* Have a clinical diagnosis of AOE in one or both ears, defined as a clinical score of at least 1 for edema (0-3 scale), 2 for overall inflammation (0-3 scale) and 1 for tenderness (absent=0, present=1).
* Be at least 18 years of age at Visit 1 (Day 1, Screening/Baseline) of either sex and any race.
* Provide written informed consent or parental assent.
* Be willing and able to follow all instructions and attend all study visits

Exclusion Criteria:

All subjects must not:

* Have known sensitivity to any component of the study medications
* Have a current infection requiring systemic antimicrobial treatment
* Have used topical or systemic pain meds on the same day as Screening/Baseline Visit 1 and for the duration of the study.
* Take any systemic (within 30 days) or otic corticosteroids (within 1 days) prior to Screening/Baseline Visit 1
* Current use of topical or systemic non-steroidal or other anti-inflammatory drugs.
* Use any topical otic treatment with alcohol, vinegar, hydrogen peroxide or other astringent medication during the course of the study or on the same day as Screening/Baseline Visit 1
* Have taken any antibiotics within 3 days prior to Visit 1
* Have signs and symptoms of AOE for > 4 weeks at Screening/Baseline Visit 1
* Have a non-intact or perforated tympanic membrane in the enrolled ear
* Have a clinical diagnosis of chronic suppurative otitis media, acute otitis media or acute otorrhea in patients with tympanostomy tubes
* Have a clinical diagnosis of malignant otitis externa
* Have overt fungal AOE
* Have a viral infection of the pinna or tympanic membrane (i.e herpes zoster)
* Have congenital abnormalities of the external auditory canal in the enrolled ear(s)
* Have obstructive bony exostoses in the enrolled ear(s)
* Have mastoid or other suppurative, non-infectious ear disorders (e.g, cholesteatoma)
* Have malignant tumors of the external auditory canal
* Have a history of otologic surgery. Surgery performed more than 1 year prior to Screening/Baseline Visit 1and limited to the tympanic membrane is allowed
* Have seborrheic dermatitis of the external auditory canal
* Have a current or prior history of immunosuppressive disorders
* Have acute or chronic renal insufficiency, hepatitis or diabetes mellitus
* Be pregnant, nursing or planning a pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-07-31 (Actual); Primary Completion 2010-07-31 (Actual); Study Completion 2010-07-31 (Actual)

PRIMARY OUTCOMES:
Overall clinical cure as defined by absence of the signs and symptoms of AOE including ear inflammation, edema, tenderness and otic discharge. | 1 year

SECONDARY OUTCOMES:
Microbiological resolution defined as elimination of pre-treatment pathogenic bacteria. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (5):
- United States (5):
  - ENT Associates of South Florida, Boynton Beach, Florida
  - Sarasota, Florida
  - Austin Ear, Nose, and Throat Clinic, Austin, Texas
  - San Antonio Ear, Nose, and Throat Research, San Antonio, Texas
  - Ear Institute of Texas, San Antonio, Texas